CLINICAL TRIAL: NCT06651047
Title: Pharmacokinetic/Pharmacodynamic Analysis of Ceftazidime/Avibactam or Cefiderocol With or Without Fosfomycin for the Treatment of Difficult To-treat Gram-negative Infections
Brief Title: PK/PD Analysis of Ceftazidime/Avibactam or Cefiderocol With or Without Fosfomycin for the Treatment of Difficult To-treat Gram-negative Infections
Acronym: PACCOF
Status: Recruiting | Type: Observational
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Maddalena Giannella, Professor, University of Bologna
Other Study IDs: PACCOF; NextGenerationEU (Other Grant/Funding Number: European Union)
Record Dates: First submitted 2024-10-15; First posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Gram Negative Infection; Antimicrobial Resistance (AMR)
Keywords: Gram-negative infection; Ceftazidime/Avibactam; Cefiderocol; Fosfomycin; Pharmacokinetics/Pharmacodynamics targets; Carbapenem-resistant Enterobacterales (CRE)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * Serum samples for PK/PD analysis
  * Serum samples for identification of new biomarkers
  * Isolated bacterial strains
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with difficult-to-treat gram-negative infection treated with CAZ/AVI or CEF, ± FOS: All patients (any age) with infection due to a difficult-to-treat Gram-negative bacteria treated with CAZ/AVI alone, CEF alone, CAZ/AVI plus FOS, or CEF plus FOS

SUMMARY:
A multicenter, national, prospective, observational pharmacological study of patients with difficult-to-treat Gram-negative infections treated with ceftazidime/avibactam (CAZ/AVI) or cefiderocol (CEF) monotherapy or combination therapy with ceftazidime/avibactam associated with fosfomycin (FOS) or cefiderocol associated with fosfomycin.

DETAILED DESCRIPTION:
Gram-negative infections, particularly those caused by Carbapenem-resistant Enterobacterales (CRE), have a dramatic impact on patient survival. Despite the introduction of new drugs in the last years have improved the outcome of patients with difficult-to-treat gram-negative infections, mortality and relapse rates are still relevant, especially in patients with high-risk sources such as pneumonia, and those in which the attainment of optimal exposure could be reduced by underlying renal disease. The use of a combination regimen in these scenarios has been proposed. However, a standardized approach to therapeutic management is still missing. To overcome this unmet clinical need, this study aims to investigate the pharmacokinetic/pharmacodynamics (PK/PD) optimization of antibiotic dosing regimens in patients with difficult-to-treat Gram-negative infections, using Therapeutic Drug Monitoring (TDM). A prompt implementation of an appropriate targeted antibiotic therapy could represent a valuable approach to improve clinical outcomes in patients with difficult-to-treat Gram-negative infections. Moreover, more information is needed in pediatric populations where ceftazidime/avibactam (CAZ/AVI) is approved only for children aged > 3 months (with the same indications as adults) and cefiderocol (CEF) is not approved. Indeed, cefiderocol is currently off-label administered in pediatric population using case-by-case dosages based on encouraging case reports.

Since several in vitro studies have highlighted the synergistic effect of fosfomycin (FOS) with different antibiotic classes, including cephalosporins such drug could be an appealing option in combination therapy for the management of difficult-to-treat gram-negative infections, both with CAZ/AVI and CEF. However, real-life prospective studies are needed to investigate the potential benefit of combination therapy on clinical outcomes and the occurrence of further resistance. Thus, the correct dose of FOS along with the type of administration (i.e., intermittent, extended, or continuous infusion) are issues to establish.

In particular, the primary aim of the study is to evaluate the probability of achieving pre-determined pharmacokinetic/pharmacodynamic (PK/PD) efficacy targets for CAZ/AVI, CEF and FOS.

Secondary objectives are:

* to evaluate the relationship between the achievement of the PK/PD target of CAZ/AVI, CEF and FOS and microbiological eradication;
* to evaluate the trend of clinical biomarkers in response to antibiotic therapy;
* to investigate the diagnostic and prognostic value of protein biomarkers.

This research is supported by EU funding within the Next Generation EU-MUR PNRR Extended Partnership initiative on Emerging Infectious Diseases (Project no. PE00000007, INF-ACT).

ELIGIBILITY:
Inclusion Criteria:

* Patients with infection due to a difficult-to-treat Gram-negative bacteria treated with CAZ/AVI alone, CEF alone, CAZ/AVI plus FOS, or CEF plus FOS (any age)
* Signature of the informed consent (for pediatric patients: parents or guardians able to provide consent)

Exclusion Criteria:

* Premature newborns
* Polymicrobial/mixed infections with the exception of cases with multiple Gram-negative bacteria susceptible to study drugs
* Continuous renal replacement therapy (CRRT) applications

Inclusion Criteria for Healthy Volunteer Subjects:

* Age ≥18 years
* Signature of the informed consent

Exclusion Criteria for Healthy Volunteer Subjects:

- Any known clinically relevant health problems

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with infection due to a difficult-to-treat Gram-negative bacteria, treated with CAZ/AVI alone, CEF alone, CAZ/AVI plus FOS, or CEF plus FOS (any age), hospitalized during the study period in the participating centers, will be screened for inclusion
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-07-09 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
PK/PD efficacy targets for study drugs | From enrollment (treatment onset) to the end of treatment (up to 7 days)
  Primary endpoint will be the proportion of patients achieving the PK/PD efficacy target. Since these drugs are widely used in clinical practice, safety is not evaluated in this study

SECONDARY OUTCOMES:
Difference in SOFA score | From day 0 (day of index positive culture) and day 7
  Difference in SOFA score (pSOFA for pediatric patients) between day 0 (day of index positive cultures) and day 7
Difference in C-Reactive Protein (CRP), Procalcitonin (PCT) and Interleukin-6 (IL-6) | From day 0 (day of index positive culture) and day 7
  Difference in C-Reactive Protein (CRP), Procalcitonin (PCT) and Interleukin-6 (IL-6) between day 0 and day 7
Identification of new protein-based biomarkers | From enrollment to the end of treatment (up to 7 days)
  * Difference in protein-based biomarkers at day 0 between study patients and a group of healthy subjects
  * Difference in protein-based biomarkers in study patients between different timepoints (from treatment onset to the end of treatment)
Microbiological eradication | From day 0 (day of index positive culture) and day 7
  Microbiological eradication defined as bacteremia clearance or negativization of index diagnostic samples within 7 days from index BC
Relapse and/or reinfection | From enrollment to the end of the follow-up at three months
  Relapse (new infection with the same pathogen emerging after treatment) and/or reinfection (new infection with a different pathogen emerging after treatment) rates at day 90
All-cause mortality | From enrollment to the end of the follow-up at three months
  All-cause mortality at day 30 and at day 90

CONTACTS AND LOCATIONS:
Locations (11):
- Italy (11):
  - Irccs Aoubo, Bologna
  - Azienda Ospedaliera di Rilievo Nazionale e di Alta Specializzazione (ARNAS) Garibaldi, Catania
  - ASST-FBF-Sacco, Milan
  - Azienda Ospedale - Università Padova, Padua
  - Istituto mediterraneo per i trapianti e terapie ad alta specializzazione (ISMETT), Palermo
  - Policlinico Umberto I, Rome
  - Policlinico Universitario Campus Bio-Medico, Rome
  - Ospedale Pediatrico Bambin Gesù, Rome
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome
  - Azienda Ospedaliero Universitaria Senese, Siena
  - Città della salute e della Scienza, Molinette, Turin

REFERENCES:
- See also: The study is enclosed in the INF-ACT research program that addresses pressing unmet needs of human emerging infectious diseases sith an One Health approach — https://www.inf-act.it/?l=EN